CLINICAL TRIAL: NCT04787861
Title: Improved Pulmonary Functions and Exercise Capacity in Children With Down Syndrome Following Motorized Movement Therapy: Comparison With Chest Physical Therapy
Brief Title: Motorized Movement Therapy & Pulmonary Functions in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, Hatem Abd Elmohsen Abdel Hamid Emara, Associate professor, Taibah University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Down Syndrome
Record Dates: First submitted 2021-02-12; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Functions; Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group treatment is identical to treatment of the study group but without a motorized movement device.Childen in this group received chest physical therapy program including positioning, breathing exercises, and postural drainage in addition to incentive spirometer training for 20 minutes, 3 times/week for 12 weeks.
  Interventions: Other: motorized movement therapy
- study group (Experimental): This group received the same program given to the control group in addition to an aerobic training regimen for 25 minutes 3 times/week for 12 weeks using a motorized movement device.
  Interventions: Other: motorized movement therapy

INTERVENTIONS:
Other: motorized movement therapy — The study group received an aerobic exercise regimen using a motorized movement therapy device 3 times /week in addition to the same traditional program used with the control group.

SUMMARY:
To investigate the effects of the addition of motorized movement therapy versus conventional chest physiotherapy alone on pulmonary functions, exercise capacity, and endurance in children with Down Syndrome

DETAILED DESCRIPTION:
To investigate the effects of the addition of motorized movement therapy versus conventional chest physiotherapy alone on pulmonary functions, exercise capacity, and endurance in children with Down Syndrome (DS). Methods: This randomized controlled study included 40 children (24 boys & 16 girls) with DS. Their ages ranged from 9 to 13 years. The control group received conventional chest physical therapy program, three sessions per week for 12 weeks. The study group received an aerobic exercise regimen using a motorized movement therapy device 3 times /week in addition to the same traditional program used with the control group. Pulmonary function tests, and six-minutes walking test were measured at baseline, after 18 sessions and after 36 sessions of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk independently
* No involvement in any physical rehabilitation program or sports activity
* Ability to understand and follow orders

Exclusion Criteria:

* Children suffering from obesity
* Severe visual and/or auditory impairment
* Congenital heart disease
* Children with musculoskeletal disorders

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in forced expiratory volume in 1st second (FEV1) | Baseline, week 6 and week 12
  FEV1 is the maximal volume of air that can be expired in 1st second of forced vital capacity maneuver using spirometry. We measured FEV1 at baseline and at end of 18 sessions (week 6) and 36 sessions (week 12).
Change from baseline in forced vital capacity (FVC) | Baseline, week 6 and week 12
  Forced vital capacity (FVC) is the maximal volume of air that can be expired while patient performs forced expiration as fast and as deep as possible using spirometry.
  We measured FVC at baseline and at end of 18 sessions (week 6) and 36 sessions (week 12).
Change from baseline in FEV1/FVC ratio | Baseline, week 6 and week 12
  FEV1/FVC is used to differentiate obstructive from restrictive patterns by spirometry. We measuredFEV1/ FVC at baseline and at end of 18 sessions (week 6) and 36 sessions (week 12).
Change from baseline in peak expiratory flow rate (PEFR). | Baseline, week 6 and week 12
  Peak expiratory flow rate (PEFR).is the maximal flow rate achieved during FVC maneuver using spirometry.
  We measured PEFR at baseline and at end of 18 sessions (week 6) and 36 sessions (week 12).
Change from baseline in maximum voluntary ventilation (MVV) | Baseline, week 6 and week 12
  maximum voluntary ventilation (MVV) is the maximal volume of air that can be moved by voluntary ventilation in 1 minute while the patient breathes deeply and rapidly for 12 to 15 seconds using spirometry.
  We measured MVV at baseline and at end of 18 sessions (week 6) and 36 sessions (week 12).

SECONDARY OUTCOMES:
Six-minutes walking test | Week 1,6 and 12
  The distance covered during of 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hatem A Emara, A.Prof, Principal Investigator — Taibah University
Locations (1):
- Medical Rehabilitation Hospital, Al Madīnah, Al Madinah Al Munawarah, Saudi Arabia

REFERENCES:
- [Background] Yoshimi K, Ueki J, Seyama K, Takizawa M, Yamaguchi S, Kitahara E, Fukazawa S, Takahama Y, Ichikawa M, Takahashi K, Fukuchi Y. Pulmonary rehabilitation program including respiratory conditioning for chronic obstructive pulmonary disease (COPD): Improved hyperinflation and expiratory flow during tidal breathing. J Thorac Dis. 2012 Jun 1;4(3):259-64. doi: 10.3978/j.issn.2072-1439.2012.03.17. PMID 22754664
- [Background] Pehlivan E, Niksarlioglu EY, Balci A, Kilic L. The Effect of Pulmonary Rehabilitation on the Physical Activity Level and General Clinical Status of Patients with Bronchiectasis. Turk Thorac J. 2019 Jan 1;20(1):30-35. doi: 10.5152/TurkThoracJ.2018.18093. PMID 30664424